CLINICAL TRIAL: NCT06150625
Title: Comparison Between Pragmatically Applied Orthopedic Manual Therapy and Dry Needling for Low Back Pain.
Brief Title: Pragmatically Applied Orthopedic Manual Therapy and Dry Needling for Low Back Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Youngstown State University (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-35
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Low Back Pain, Mechanical
Keywords: Low back pain, manual therapy, dry needling
MeSH Terms: conditions — Low Back Pain | interventions — Dry Needling; Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: The outcome assessor needing access to REDcap will be blinded the treatment group. The clinician providing treatment will be blinded to outcomes.
Who Masked: Outcomes Assessor
Masking Description: All data will be collected through REDcap. The treating therapist will have no knowledge pertaining to the outcomes being collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Orthopedic Manual Therapy (Active Comparator): Participants randomized to this arm will receive clinician-selected orthopedic manual therapy targeting the joints of the low back. Selected techniques can involve joint mobilizations or spinal manipulation. The dosage parameters will be determined by the clinician.
  Patient Education Patients will receive education regarding their low back pain, advice to stay active, proper performance of their home exercise program.
  Home exercise program The program will consist of 10 exercises which the clinician will select 5 they feel would be most beneficial to the patient. These can include aerobic, general strengthening, directional preference, or neural self-mobilizations.
  Interventions: Other: Orthopedic Manaual Therapy; Other: Home exercise program; Other: Patient education
- Dry Needling (Active Comparator): Participants randomized to this arm will receive dry needling to the low back and lower extremity while being applied based on clinician-selected areas of symptomatic soft tissue. The dosage parameters will be determined by the clinician.
  Patient Education Patients will receive education regarding their low back pain, advice to stay active, proper performance of their home exercise program.
  Home exercise program The program will consist of 10 exercises which the clinician will select 5 they feel would be most beneficial to the patient. These can include aerobic, general strengthening, directional preference, or neural self-mobilizations.
  Interventions: Other: Dry Needling; Other: Home exercise program; Other: Patient education
- Orthopedic Manual Therapy and Dry needling (Experimental): Participants randomized to this arm will receive dry needling to the lumbar spine and lower extremity based on clinician-selected areas of symptomatic soft-tissue and or orthopedic manual therapy targeting the joints of the low back.
  Patient Education Patients will receive education regarding their low back pain, advice to stay active, proper performance of their home exercise program.
  Home exercise program The program will consist of 10 exercises which the clinician will select 5 they feel would be most beneficial to the patient. These can include aerobic, general strengthening, directional preference, or neural self-mobilizations.
  Interventions: Other: Orthopedic Manaual Therapy; Other: Dry Needling; Other: Home exercise program; Other: Patient education

INTERVENTIONS:
Other: Orthopedic Manaual Therapy — Can include either spinal mobilizations or spinal manipulation therapy targeting the stiff or symptomatic level of the lumbar spine. Various types of mobilization or manipulation may be used based on the therapists clinical reasoning. The therapist will determine which technique and dosage parameters for each subject based on individual patient clinical data. Common mobilizations techniques involve gently and repeatedly applying pressure over different parts of the patient's spine that is associated with their symptoms. For a manipulation, the patient will be positioned in side-lying position. The therapist will then position the patient further to target the symptomatic level. The patient is asked to take a deep breathe in and out. The therapist will slowly add pressure through the trunk and apply a fast but small thrust motion toward the table.
  Arms: Orthopedic Manual Therapy; Orthopedic Manual Therapy and Dry needling
Other: Dry Needling — dry needling both sides of the symptomatic level(s) of the lumbar spine as well as needling other areas in the lower extremity and pelvis based on the results of their clinical evaluation and/or the subjects presenting symptoms. Dry needling involves the insertion of a monofilament needle (nothing is injected) into symptomatic soft tissue. The therapist will determine which technique and dosage parameters for each subject based on individual patient clinical data.
  Arms: Dry Needling; Orthopedic Manual Therapy and Dry needling
Other: Home exercise program — 5 exercises will be selected from 10 options intended to reinforce the improvements made from treatment.
Other: Patient education — Patient education on the low back condition, advice to stay active, and home exercise performance.

SUMMARY:
Both orthopedic manual therapy (OMT) and dry needling (DN) have been shown to be effective at reducing pain and disability for individuals with low back pain (LBP). It is unclear if one intervention, or in combination with one another, is more effective. The purpose of this randomized clinical trial is to determine the clinical effectiveness of OMT or DN alone compared with combined OMT + DN on pain and disability for patients with LBP. Both within and between group effects will be presented.

Patient factors such as; generalized anxiety disorder, depression, fear-avoidance behaviors, pain catastrophizing, and sleep-quality have negatively correlated with pain and disability outcomes in patients experiencing chronic LBP. Moreover, sleep deprivation and pain related fear of movement functionally can change a person's pain inhibitory pathways leading to hyeralgesia. These factors have been individually analyzed regarding their effects on pain related outcomes, which limits our understanding of how clustering patient factors might affect recovery. A secondary aim will involve determining the relationship between patient factors and clinical outcomes for individuals with LBP who receive DN and/or manual therapy.

DETAILED DESCRIPTION:
Low back pain (LBP) is a common disorder, (GBD,2016) placing a tremendous financial burden on the health care and occupational systems. (Freburg,2009) The etiology and influences to chronic LBP remains unknown due to multiple interacting factors involving pain, disability, psychosocial, and psychological factors. While the search for effective therapies has been ongoing in clinical trials, the optimal management strategies remain elusive due to inconsistent findings in randomized clinical trials (RCT) and systematic reviews. (Bussieres,2018; Coulter, 2018;Kamper, 2015)

Orthopedic manual therapy is routinely used to assist patients with LBP manage their symptoms. (George, 2021) Mechanisms identified in pre-clinical studies involve local, segmental, and systemic neurophysiological changes helping reduce pain.(Bialosky,2018) Two popular forms of orthopedic manual therapy are spinal manipulation/mobilization therapy and dry needling (DN). While these treatments share mechanisms of action, DN also creates a physiological lesion resulting in mechanical disruption of connective tissue to deeper structures. Clinical Practice Guidelines recommend both OMT and DN be incorporated as part of a multimodal treatment plan.(George,2021) It is unknown if these treatments combined produce larger treatment effects than when they are applied individually. While this treatment combination has been investigated for other musculoskeletal conditions (Dunning, 2021a; Dunning, 2021b; González-Iglesias,2013; Gattie, 2021), it has not been studied for LBP.

Patient Factors that Influence Outcomes Patient factors such as generalized anxiety disorder, depression, fear-avoidance behaviors, pain catastrophizing, and sleep-quality have negatively correlated with pain and disability outcomes in patients experiencing chronic LBP. (Alhowimel,2018) A recent multimodal metanalysis involving patients with depressive/anxiety disorders with chronic pain observed disorder specific neurological changes on functional MRI, exploiting neuro-behavioral mechanisms. (Brandl 2022) Moreover, sleep deprivation and pain related fear of movement functionally can change a person's pain inhibitory pathways leading to hyeralgesia. (Finan 2013; Meier, 2017) These factors have been individually analyzed regarding their effects on pain related outcomes, which limits our understanding of how clustering patient factors might affect recovery. We hypothesize that certain combinations of patient factors will correlate with those patients with chronic LBP who were less likely to experience a clinically meaningful change in pain and disability.

Statement of the Problems

Problem 1: The most effective conservative management strategies for patients with LBP remains unknown. Manual therapy is routinely used in clinical practice and recommended in Clinical Practice Guidelines, including OMT and DN. It is unknown if a pragmatically applied OMT combined with DN produces larger treatment effects than a pragmatically applied SMT alone for patients with LBP.

Problem 2: Patient factors such as psychological and psychosocial factors, patient recovery expectations, and patient treatment preferences have all demonstrated the ability to influence clinical outcomes in patients with LBP. Currently it is not understood how the presence of multiple patient variables combine to interact with patient outcomes.

Purpose Statement The purpose of this randomized clinical trial is to determine the clinical effectiveness of OMT or DN alone compared with OMT and DN on pain and disability for patients with LBP. Both within and between group effects will be presented. Our hypothesis is that individuals treated with both OMT and DN will experience greater changes in pain and disability compared with those who receive either treatment individually. We also anticipate the presence of patient factors known to influence pain will negatively correlate with patient outcomes and certain combinations of these patient factors may have a stronger influence on clinical outcomes.

Statement of Research Objectives

Specific Aim 1: Determine the comparative effectiveness of pragmatically applied OMT with DN compared to OMT or DN alone for patients with LBP and disability.

Specific Aim 2: Determine the relationship between patient factors and clinical outcomes for individuals with LBP who receive DN and/or OMT.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years of age or older, present with LBP and a pain score of > or = 3/10

Exclusion Criteria:

* Patients will be excluded if they present with a contraindication to either treatment (malignancy, fracture, myelopathy, osteoporosis, etc.), have a prior surgical history involving the lumbar spine, present with spinal nerve root compression (2 or more neurological findings that includes myotome weakness, dermatomal sensory loss, and/or deep tendon reflexive changes), are seeking litigation, or are receiving other forms of conservative care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
PROMIS-29.2 | Baseline, 1 week, 1 month, and 6 months
  Questionnaire that assesses 7 domains with 4 questions with an additional pain intensity numeric rating scale (NPRS). The PROMIS measures have been tested and validated in large reference populations making them suitable for research on different conditions.

SECONDARY OUTCOMES:
Global Rating of Change | 1 week, 1 month, and 6 months
  Questionnaire that assesses the global degree of change the patient perceives since the start of care.
  The patient rates their change from 0 (no change) to +7 (A Very Great Deal Better) to -7 (A Very Great Deal Worse)
Global Rating of Change for Medication Intake | 1 week, 1 month, and 6 months
  Questionnaire that assesses the global degree of change in pain medication the patient experienced since the start of care. The patient rates their change in medications from 0 (no change) to +7 (A Very Great Deal Less) to -7 (A Very Great Deal More)
Health Care Utilization | 6 months
  Patients will report any providers they had to see after the completion of the study to 6 months for their low back problem.

OTHER OUTCOMES:
Patient Treatment Preference | Baseline
  The patient rates their preference for treatment between dry needling, orthopedic manual threrapy, or both.
Clinician Treatment Preference | Baseline
  The clinician rates their preference for treatment between dry needling, orthopedic manual threrapy, or both.
Credibility Expectancy Questionnaire | Baseline
  Scale for measuring treatment expectancy and rationale credibility for use in clinical outcome studies.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rubinstein SM, de Zoete A, van Middelkoop M, Assendelft WJJ, de Boer MR, van Tulder MW. Benefits and harms of spinal manipulative therapy for the treatment of chronic low back pain: systematic review and meta-analysis of randomised controlled trials. BMJ. 2019 Mar 13;364:l689. doi: 10.1136/bmj.l689. PMID 30867144
- [Background] Hu HT, Gao H, Ma RJ, Zhao XF, Tian HF, Li L. Is dry needling effective for low back pain?: A systematic review and PRISMA-compliant meta-analysis. Medicine (Baltimore). 2018 Jun;97(26):e11225. doi: 10.1097/MD.0000000000011225. PMID 29952980
- [Background] Corp N, Mansell G, Stynes S, Wynne-Jones G, Morso L, Hill JC, van der Windt DA. Evidence-based treatment recommendations for neck and low back pain across Europe: A systematic review of guidelines. Eur J Pain. 2021 Feb;25(2):275-295. doi: 10.1002/ejp.1679. Epub 2020 Nov 12. PMID 33064878
- [Background] Owen PJ, Miller CT, Mundell NL, Verswijveren SJJM, Tagliaferri SD, Brisby H, Bowe SJ, Belavy DL. Which specific modes of exercise training are most effective for treating low back pain? Network meta-analysis. Br J Sports Med. 2020 Nov;54(21):1279-1287. doi: 10.1136/bjsports-2019-100886. Epub 2019 Oct 30. PMID 31666220